CLINICAL TRIAL: NCT06363799
Title: Osteopathic Protocol for Insomnia in College Students: RCT
Brief Title: Osteopathic Protocol for Insomnia in College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Prinicipal Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OST1_010
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Insomnia
Keywords: CV4; Diaphragmatic breathing; Insomnia; Osteopathy; College Students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4th ventricle compression technique (Experimental): Experimental:
  4th ventricle compression technique
  Interventions: Other: 4th ventricle compression technique
- Diaphragmatic breathing technique (Experimental): Experimental:
  Diaphragmatic breathing technique
  Interventions: Other: Diaphragmatic breathing technique
- Sham Tecnhique (Placebo Comparator): Placebo Comparator:
  Sham Technique
  Interventions: Other: Sham Technique

INTERVENTIONS:
Other: 4th ventricle compression technique — For the CV4 the mediator's hands assume a specific position: one on top of the other, with the tips of the thumbs joined together in a "V" shape, positioned approximately on the process spinous between the patient's second and third cervical vertebrae, pointing downwards.
  Arms: 4th ventricle compression technique
Other: Sham Technique — The participant is instructed to lie down in the supine position while the mediator assumes a position at the head of the table and places their hands on the participant's shoulders. This technique is performed for 5 minutes.
  Arms: Sham Tecnhique
Other: Diaphragmatic breathing technique — For the diaphragmatic breathing the participant will place one hand on their chest and the other over their abdomen. Both of their hands will be overlapped by the mediator's, so it is easier to feel the correct breathing movements to be performed.
  Arms: Diaphragmatic breathing technique

SUMMARY:
In this randomized controlled experimental trial, it is aimed to determine the effectiveness of an osteopathic protocol treatment for insomnia in college students. In this study, will be used the Compression of 4th ventricle (CV4) and the diaphragmatic breathing technique.

DETAILED DESCRIPTION:
Insomnia is a sleep disorder defined by persistent difficulty in initiating, maintaining or consolidating sleep. It can also be defined by early morning awakenings or having a dissatisfied sleep quality, even if you have plenty of time and a suitable environment to a restful sleep. This difficulty sleeping must be experienced at least 3 nights per week, for 3 consecutive months. This can often lead to symptoms such as fatigue, irritability and difficulty concentrating during the day.

Both compression of 4th ventricle and diaphragmatic techniques have been proven to help lower the tone of the sympathetic nervous system, restoring a normal respiratory mechanism.

It is anticipated that the combination of 4th ventricle technique and diaphragmatic breathing may result in a significant reduction in insomnia symptoms, providing study participants with a notable improvement in the quality of sleep and, therefore, in their general well-being.

ELIGIBILITY:
Inclusion Criteria:

* being a college student
* insomnia presence
* willingness to complete a full study period
* understanding and acceptance of the study procedures
* willingness to refrain from other intervention during the study period
* availability to keep a diary (sleep and mood throughout the day)

Exclusion Criteria:

* having suffered a stroke or aneurysm
* hypertension
* fractured the base of the skull
* pregnancy
* active insomnia treatment
* participation in other simultaneous studies
* regular use of sleep medication
* have participated in complementary therapies for insomnia recently

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline insomnia episodes and symptoms through Pittsburgh questionnaire score | One month after the first intervention
  The insomnia episodes and symptoms are measured using the Pittsburgh questionnaire and it will be applied one month after the first intervention. It is expected that the Pittsburgh score decreases after the intervention is done. A Pittsburgh score higher than 5 is considered to be coincident with a bad sleeping quality. A Pittsburgh score lower than 5 is considered to be coincident with a good sleeping quality. This score goes up to 21 points.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior da Saúde do Porto

REFERENCES:
- [Background] Bordoni B, Escher AR Jr. Osteopathic Principles: The Inspiration of Every Science Is Its Change. Cureus. 2021 Jan 4;13(1):e12478. doi: 10.7759/cureus.12478. PMID 33425556
- [Background] Cardoso-de-Mello-E-Mello-Ribeiro AP, Rodriguez-Blanco C, Riquelme-Agullo I, Heredia-Rizo AM, Ricard F, Oliva-Pascual-Vaca A. Effects of the Fourth Ventricle Compression in the Regulation of the Autonomic Nervous System: A Randomized Control Trial. Evid Based Complement Alternat Med. 2015;2015:148285. doi: 10.1155/2015/148285. Epub 2015 Jun 14. PMID 26199632
- [Background] Chen YF, Huang XY, Chien CH, Cheng JF. The Effectiveness of Diaphragmatic Breathing Relaxation Training for Reducing Anxiety. Perspect Psychiatr Care. 2017 Oct;53(4):329-336. doi: 10.1111/ppc.12184. Epub 2016 Aug 23. PMID 27553981
- [Background] Consolo, K., Fusner, S., & Staib, S. (3 de Outubro de 2008). Effects of diaphragmatic breathing on stress levels of nursing students. pp. 67-71.
- [Background] DiGiovanna , E., Schiowitz, S., & Dowling, D. (2020). An Osteopathic Approach to Diagnosis and Treatment, Fourth Edition. Lippincott Williams & Wilrins.
- [Background] Homistek, C., & Doty, H. (2021). Insomnia Diagnosis and Management: An Osteopathic Approach. Osteopathic Family Physician, 31-36.
- [Background] Lande RG, Gragnani C. Nonpharmacologic approaches to the management of insomnia. J Am Osteopath Assoc. 2010 Dec;110(12):695-701. PMID 21178150
- [Background] Liem, T., McPartland, J., & Skinner, E. (2005). Cranial Osteopathy - Principles and Practice. Elsevier Health Sciences.
- [Background] Liu D, Kahathuduwa C, Vazsonyi AT. The Pittsburgh Sleep Quality Index (PSQI): Psychometric and clinical risk score applications among college students. Psychol Assess. 2021 Sep;33(9):816-826. doi: 10.1037/pas0001027. Epub 2021 May 20. PMID 34014747
- [Background] Manzar MD, BaHammam AS, Hameed UA, Spence DW, Pandi-Perumal SR, Moscovitch A, Streiner DL. Dimensionality of the Pittsburgh Sleep Quality Index: a systematic review. Health Qual Life Outcomes. 2018 May 9;16(1):89. doi: 10.1186/s12955-018-0915-x. PMID 29743066
- [Background] McCarley RW. Neurobiology of REM and NREM sleep. Sleep Med. 2007 Jun;8(4):302-30. doi: 10.1016/j.sleep.2007.03.005. Epub 2007 Apr 30. PMID 17468046
- [Background] Milnes, K., & Moran, R. (17 de Janeiro de 2007). Physiological effects of a CV4 cranial osteopathic technique on autonomic nervous system function: A preliminary investigation. pp. 8-17.
- [Background] Morin M., C., Beaulieu-Bonneau, S., & Cheung, J. (2019). Treatment of Insomnia. Em Handbook of Sleep Disorders in Medical Conditions. Elsevier.
- [Background] Pacheco, D., & Dimitriu, A. (2022). Symptoms of Insomnia.
- [Background] Zitser J, Allen IE, Falgas N, Le MM, Neylan TC, Kramer JH, Walsh CM. Pittsburgh Sleep Quality Index (PSQI) responses are modulated by total sleep time and wake after sleep onset in healthy older adults. PLoS One. 2022 Jun 24;17(6):e0270095. doi: 10.1371/journal.pone.0270095. eCollection 2022. PMID 35749529